CLINICAL TRIAL: NCT06721559
Title: Empower@Home: Community Implementation for Older Adults With Ambulatory Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00259594; 90IFRE0097 (Other Grant/Funding Number: ACL/NIDILRR)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Depression
Keywords: Cognitive behavioral therapy; Older adults; Internet-based intervention; Depression; Social isolation
MeSH Terms: conditions — Depression; Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding interventionalists and participants is not possible, given the nature of the intervention. However, assessment staff will be blinded when possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empower@Home supported by aging service providers (Experimental): Participants will be provided with access to a 9-session online program called Empower@Home, a self-help intervention based on cognitive behavioral therapy principles. The intervention has three components: 9 interactive self-paced online sessions, printed workbook that goes along the online sessions for exercises and homework, and telephone coaching by a trained staff from a social service agency serving older adults. Participants will have up to 12 weeks to try to complete the program with the support of a trained coach.
  Interventions: Behavioral: Empower@Home: An online cognitive-behavioral therapy self-care program for geriatric depression
- Attention call with friendly visitors (Other): Participants will receive enhanced care as usual, including care as usual from their social service provider and a psycho-educational handout. In addition, they will receive telephone friendly calls from a research staff every other week to mimic the human interactions provided by coaches in the experimental group.
  Interventions: Other: Telephone friendly visits

INTERVENTIONS:
Behavioral: Empower@Home: An online cognitive-behavioral therapy self-care program for geriatric depression — Empower@Home is an online self-help intervention based on cognitive behavioral therapy principles designed to treat depressive symptoms in older adults. The intervention has three components: 9 interactive self-paced online sessions, printed workbook that goes along the online sessions for exercises and homework, and telephone coaching by a trained staff from a social service agency serving older adults. The online sessions contain entertainment elements in the form of a character-driven story of a homebound older adults, video-based psycho-educational content, voice-over instructions, interactive exercises, and weekly home practice assignments.
  Arms: Empower@Home supported by aging service providers
Other: Telephone friendly visits — Participants in the waitlist control group will receive attention control through biweekly telephone-friendly visitors. Trained project staff will call participants to provide companionship, emotional support, and a friendly conversation. In addition, the callers will conduct a biweekly assessment of depressive symptoms using the patient health questionnaire (PHQ-9), to mirror the biweekly in-app PHQ-9 assessments with the experimental group.
  Arms: Attention call with friendly visitors

SUMMARY:
This study is a randomized Type I hybrid effectiveness-implementation trial aimed at evaluating the effectiveness of Empower@Home, an internet-delivered cognitive-behavioral therapy (CBT) program supported by social service providers, in comparison to enhanced usual care for depression in older adults with ambulatory disabilities. A total of 64 participants with ambulatory disabilities will be randomly assigned to either the treatment group (Empower@Home) or the control group (enhanced usual care) in a 1:1 allocation ratio.

This project addresses the following research questions:

1. Does the intervention affect individuals' lives in the following expected areas?

   1. Does participation in the intervention lead to greater improvement in depressive symptoms than enhanced care as usual?
   2. Does participation in the intervention lead to greater improvement in social engagement and activities than enhanced care as usual?
   3. Is the intervention's primary effect mediated by CBT-related (e.g., CBT skills acquisition, cognitive distortions, and behavioral activation), engagement-related (e.g., character or storyline relatedness), and coach-related factors (e.g., therapeutic alliance)?
2. How is the intervention being adopted? What are the barriers and facilitators encountered during the implementation process?

DETAILED DESCRIPTION:
This study is a randomized Type I hybrid effectiveness-implementation trial designed to evaluate the clinical effectiveness and implementation process of Empower@Home, an internet-delivered cognitive-behavioral therapy (CBT) program tailored for homebound older adults with depressive symptoms. The trial compares Empower@Home, supported by aging service providers, to an enhanced usual care condition. The study involves 64 participants with ambulatory disabilities who will be randomly assigned to either the treatment or control group.

Rationale: Depression is a significant public health concern among homebound older adults, with approximately 50% experiencing clinically significant depressive symptoms and 14% facing major depression-rates significantly higher than those of non-homebound counterparts. Homebound older adults often encounter barriers to accessing traditional mental health services, including physical disabilities, socioeconomic disadvantages, and racial or ethnic minority status. Empower@Home addresses these challenges by leveraging the existing workforce of aging service providers to support digital mental health interventions (DMHIs).

Intervention: Empower@Home is a nine-session, computerized CBT program enhanced with entertainment elements to increase engagement. The program is specifically designed for homebound older adults, incorporating age-relevant examples and a simplified user interface. It includes features such as a character-driven storyline, short videos, and interactive exercises to facilitate learning and engagement. The program is supported by lay coaches-aging service providers trained to offer weekly support calls, enhancing program adherence and personalization.

This project addresses the following research questions:

1. Does the intervention affect individuals' lives in the following expected areas?

   1. Does participation in the intervention lead to greater improvement in depressive symptoms than enhanced care as usual?
   2. Does participation in the intervention lead to greater improvement in social engagement and activities than enhanced care as usual?
   3. Is the intervention's primary effect mediated by CBT-related (e.g., CBT skills acquisition, cognitive distortions, and behavioral activation), engagement-related (e.g., character or storyline relatedness), and coach-related factors (e.g., therapeutic alliance)?
2. How is the intervention being adopted? What are the barriers and facilitators encountered during the implementation process?

Study Design: Participants will be recruited from an aging service agencies that serve as implementation sites. Participants will undergo remote assessments via phone at baseline, post-intervention, and a follow-up at 24 weeks.

Expected Outcomes: The study is expected to demonstrate that Empower@Home, when supported by aging service providers, is more effective than usual care and friendly calls in reducing depressive symptoms and improving social engagement and activities participation. Additionally, the findings will provide valuable insights into the barriers and facilitators to implementing DMHIs in community settings, offering guidance for future scalability and sustainability of such interventions.

Innovation: Empower@Home integrates user-centered design principles, community participatory research, and innovative engagement strategies, such as character-driven storytelling, to enhance user experience and therapeutic outcomes. The use of aging service providers as lay coaches not only addresses the shortage of mental health professionals but also aligns with the existing infrastructure of aging services, making the program highly scalable and sustainable.

This trial will contribute significantly to the growing body of evidence on the effectiveness of DMHIs in real-world settings and inform strategies for broader implementation within community-based aging and disability services.

ELIGIBILITY:
Inclusion Criteria:

* (1) be receiving or eligible to receive services at the recruitment sites
* (2) read and speak English
* (3) be at least 50 years old
* (4) have at least mild depressive symptoms at screening (≥ 5 on the Patient Health Questionnaire-9 [PHQ-9]).
* (5) Participants who are NOT currently receiving outside therapy must agree NOT to start outside therapy during study participation. Participants who are currently receiving outside therapy must agree NOT to increase their outside therapy frequency during study participation.
* (6) have mobility limitations based on self-reported limitations in 10 mobility related questions (e.g., difficulty climbing stairs or walking)

Exclusion Criteria:

* (1) probable dementia based on the Blessed Orientation and Memory Scale.
* (2) moderate or high risk of suicide based on the 6-item Columbia-Suicide Severity Rating Scale
* (3) a terminal illness with less than six months to live or unstable physical health conditions based on self-report
* (4) a diagnosis of a psychotic disorder like schizophrenia or bipolar disorder based on self-report and medical chart review
* (5) severe vision impairment based on self-report (i.e., legally blind)
* (6) current substance use disorders or receiving substance use treatment.
* (7) currently receiving outside therapy more frequently than once a month or have started a new therapy treatment less than 3 months ago

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline to follow-up assessments at 12 and 24 weeks
  Change in 9 item standardized measures of depressive symptom severity. PHQ-9 score ranges from 0 to 27, with a higher score indicating more severe symptoms.
Change in Social Engagement and Activities Questionnaire (SEAQ) | Change from Baseline to follow-up assessments at 12 and 24 weeks
  Change in 10 item standardized measures of participation in social activities and community participation. The total scores range from 0 to 50, and a higher score suggesting a higher level of participation.

SECONDARY OUTCOMES:
Change in Duke Social Support Index (DSSI)-10 | Change from Baseline to follow-up assessments at 12 and 24 weeks
  Change in 10 item standardized measure for social interaction and satisfaction with social support. Total score ranges from 10 to 30, higher score means higher social support.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared through ICPSR, in compliance with NIDILRR funding requirements. The data will be available to qualified researchers following appropriate data use agreements. All quantitatively collected, non-identifying IPD, along with data dictionaries will be deposited to ICPSR.
Supporting Information: ICF
Time Frame: Within one year of study conclusion
Access Criteria: Apply through ICPSR
URL: https://www.icpsr.umich.edu/web/datamanagement/cms/5292

REFERENCES:
- See also: Intervention website — https://empower-at-home.com/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT06721559/ICF_001.pdf